CLINICAL TRIAL: NCT07392684
Title: Optimisation of the Blood Culture Pathway Utilising Behaviour Change
Status: Recruiting | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24/043/GHT
Record Dates: First submitted 2025-09-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Microbiology; Blood Culture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Staff members that collect adult blood cultures within the Trust

SUMMARY:
Blood culture (BC) is the gold standard for the definitive diagnosis of bacteraemia, providing the opportunity to recover and identify the causative organism, and optimize subsequent antimicrobial treatment. Detection of bacteraemia is critical for the management of sepsis. This study aims to examine the performance of the blood culture pathway in Gloucestershire Hospitals Trust using data analysis, questionnaires and focus groups. . Information collected will be used to design interventions that could be used to optimise the blood culture pathway

DETAILED DESCRIPTION:
Retrospective data collection relating to the blood volume collected and time to incubation of adult blood culture sets (adult sets comprises of both aerobic and anaerobic blood culture bottle) received in the microbiology laboratory, between February 2023 and April 2024. These samples are routinely collected as standard of care and not for the purpose of this research.

Staff members that collect adult blood cultures within the Trust (nurses, Physician's associates and doctors) will be invited to volunteer for the study. Staff members will participate by completing the questionnaire and/or attending focus groups.

ELIGIBILITY:
Inclusion Criteria:

Secondary data:

- adult blood culture sets received in the microbiology laboratory, between February 2023 and April 2024.

Staff member participants

- Staff members that collect adult blood cultures within the Trust

Exclusion Criteria:

Secondary data:

* paediatric blood culture samples
* samples where volume, collection and/or time to incubation data are not recorded on laboratory system and/or blood culture analyser

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary data: adult blood culture sets received in the microbiology laboratory, between February 2023 and April 2024.
  Staff member participants: Staff members that collect adult blood cultures within the Trust
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Compliance to optimal blood culture (BC) vol (8-10 mls per bottle). | Retrospective data collection from period February 2023 to April 2024.
  Volume of blood cultures measured in ml.
Compliance to 4- hour time target to incubation of blood culture from collection. | Retrospective data collection from period February 2023 to April 2024
  Time taken from collection of blood culture to incubation in the laboratory, recorded in hours and minutes
Time from collection of blood cultures to targeted antibiotics, hours and minutes | Retrospective data collection from period February 2023 to April 2024.
  Measurement of time (hours, minutes) from time of blood culture collection to time of targeted antibiotic prescribing
Staff experiences related to taking blood cultures | Approximately 10 minutes to complete electronic questionnaire. Attendance at single FOCUS group at agreed time.
  Staff experiences using questionnaires and focus group discussions exploring facilitators and barriers relating to blood culture collection . Staff members will participate by completing the questionnaire and/or attending focus groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Gloucestershire Royal Hospital, Gloucester, Gloucestershire, United Kingdom